CLINICAL TRIAL: NCT00322192
Title: The Effects of Functional Strength Training on Weakness and Function of the Lower Limb After Stroke
Brief Title: Evaluation of Whether Functional Strength Training Can Enhance Recovery of Mobility After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: The Health Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Health Foundation 224/1960; Health Foundation 224/1960
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2006-05

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; Physical Therapy
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Behavioral: Conventional UK Physical therapy
Behavioral: Increased intensity of UK conventional physical therapy
Behavioral: UK conventional physical therapy plus functional strength training

SUMMARY:
The purpose of this study is to test the hypothesis that adding functional strength training to UK conventional therapy improves muscle function and walking than either UK conventional therapy alone or increased intensity of UK conventional therapy

DETAILED DESCRIPTION:
Neuromuscular weakness occurs frequently after stroke and the processes underlying recovery are still poorly understood. Accepted practice in UK physiotherapy is to avoid training of muscle strength after stroke but there is preliminary evidence that it might be effective.

An observer-blind randomised clinical trial. Subjects will be within 3 months of first stroke with some voluntary movement in the paretic lower limb. A power calculation estimated the sample size as 300. Research Physiotherapists, blinded to measurement, will recruit subjects, allocate subjects to one of the three intervention groups using sequentially numbered sealed envelopes containing previously randomised allocated intervention cards and provide interventions. The Research Assessors, blinded to intervention allocation will undertake all measurements. Conventional therapy (control) will be provided as normal for the clinical setting, the additional conventional therapy (experimental 1) or functional strength training (experimental 2) will be provided for one hour, four times a week, for six weeks. Subjects in the two experimental groups will also receive the conventional therapy standard in their clinical setting. Blinded measurement will be made before randomisation, at the end of intervention and 12-weeks thereafter. Primary outcomes are maximum torque around the knee joint, and gait velocity. The secondary outcomes include movement analysis, functional ability, corticospinal transmission (transcranial magnetic stimulation) and health related quality of life (Euroqol). The primary analysis will be analysis of covariance. A multiple comparison procedure (Gabriel's test) will be used to compare each pair of treatments. Euroqol data will be used to estimate the relative costs of the interventions and to calculate the incremental cost per QUALY gained. Every effort will be made to invite patients for assessment at outcome and follow-up even if they have withdrawn from therapy to allow the intention-to-treat principle to be applied.

ELIGIBILITY:
Inclusion Criteria:

Subjects in this study will:

* be aged over 50 years.
* be between one week and three months after stroke when recruited to the study;
* have been independently mobile indoors, with or without aids, before the stroke;
* have some voluntary movement in the paretic lower limb i.e. score above 28/100 on the lower limb section of the Motricity Index43;
* demonstrate adequate orientation and communication (be able to complete a one-stage command using the non-paretic upper limb e.g. point at the ceiling).

In addition those who agree to participate in TMS measurement will have no contraindications to TMS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Maximum torque around the knee joint
gait velocity

SECONDARY OUTCOMES:
Modified Rivermead Mobility Index
Lower limb kinematics during standing up
Lower limb kinematics during sitting down
Lower limb kinematics during walking
timing and pattern of muscle activation during functional activity
EuroQuol for health related quality of life
Transmission in the corticospinal pathways for suitable subjects who provide additional written informed consent for TMS

CONTACTS AND LOCATIONS:
Overall Officials: Valerie M Pomeroy, PhD, Study Chair — St George's University London, UK; Emma V Cooke, MSc, Principal Investigator — St George's University London, UK; Raymond C Tallis, FMedSci, Study Director — University of Manchester
Locations (4):
- United Kingdom (4):
  - St George's Hospital NHS Trust, London, London
  - Epsom and St Helier NHS Trust, Carshalton, Surrey
  - Ashford and St Peter's Hospitals NHS Trust, Chertsey, Surrey
  - Mayday University Hospital NHS Trust, Thornton Heath, Surrey

REFERENCES:
- [Derived] Kerr A, Clark A, Cooke EV, Rowe P, Pomeroy VM. Functional strength training and movement performance therapy produce analogous improvement in sit-to-stand early after stroke: early-phase randomised controlled trial. Physiotherapy. 2017 Sep;103(3):259-265. doi: 10.1016/j.physio.2015.12.006. Epub 2016 Feb 11. PMID 27107979